CLINICAL TRIAL: NCT03951181
Title: A Single-Arm Feasibility Study of the Life-Style Exercise and Activity Package for People Living With Progressive Multiple Sclerosis
Brief Title: Life-Style Exercise and Activity Package for People Living With Progressive MS
Acronym: LEAP-MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SPON1666-18
Record Dates: First submitted 2019-05-07; First posted 2019-05-15 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LEAP-MS Intervention (Experimental): This is a single arm study.
  Interventions: Behavioral: LEAP-MS

INTERVENTIONS:
Behavioral: LEAP-MS — The LEAP-MS intervention is a co-produced, digital interactive education and activity tool, specifically developed for PwPMS. The tool includes multimedia education about being active with PMS, tailored physical activity ideas and interactive functions enabling the development of personalised activity programmes, goal setting and activity logs. The digital tool works in conjunction with support from trained physiotherapists. The feasibility study will evaluate how the LEAP-MS intervention can be used in practice.

SUMMARY:
The investigators know that many people with multiple sclerosis (MS) require support to remain physically active and often do not receive any or enough support. This is particularly the case for People with Progressive MS (PwPMS) with moderate to severe disability - those who require assistance to mobilise (i.e. using a stick, frame or wheelchair) and/or have other MS related symptoms such as fatigue and difficulties remembering.

In Phase 1 of the LEAP-MS study the investigators collected information about the barriers to and facilitators of physical activity (PA) that PwPMS experience, their current levels and type of physical activity and their perceptions of the role physical activity plays in managing MS symptoms from both them and their families - or people that support them. This provided important information about why physical activity might be important for PwPMS, the challenges they face in doing physical activity or accessing it, and ways which they have found to overcome any barriers. The investigators also collected information from physiotherapists and other health care professionals who specialise in treating people with MS, about their understanding of self-management and their needs for training about using self-management approaches with PwPMS. The investigators used this information to co-produce (with the involvement of PwPMS patients and physiotherapists/healthcare professionals) a personalised intervention; Life-style, exercise and activity package for people living with progressive multiple sclerosis (LEAP-MS) to facilitate on-going physical activity for people with PwPMS and a training package about self-management with PwPMS for physiotherapists.

In this feasibility study the investigators will evaluate the acceptability of the LEAP-MS intervention. The investigators will also evaluate feasibility of conducting a future trial of the intervention in terms of recruitment, retention, adherence (usage), outcome measures and safety evaluation and establishing fidelity of intervention delivery.

DETAILED DESCRIPTION:
Primary objectives. The primary objective is to establish the feasibility, acceptability and fidelity and safety of the LEAP-MS intervention for PwPMS and physiotherapists.

Secondary objectives. The secondary objectives are to validate the proposed intervention logic model through both qualitative assessment of intervention processes and descriptive evaluation of potential outcomes.

Study design and setting. This is a single arm feasibility study with an embedded process evaluation.

Study Intervention. The LEAP-MS intervention is a co-produced, digital interactive education and activity tool, specifically developed for PwPMS. The tool includes multimedia education about being active with PMS, tailored physical activity ideas and interactive functions enabling the development of personalised activity programmes, goal setting and activity logs. The digital tool works in conjunction with support from trained physiotherapists. The feasibility study will evaluate how the LEAP-MS intervention can be used in practice.

Patient participant study procedure. The investigators aim to recruit 21 PwPMS to participate in the LEAP-MS feasibility study. Patients will self refer to the LEAP-MS website.

Training physiotherapists. Physiotherapists will be trained on how to deliver self-management support to the participants. This training will have been developed following the information collected from physiotherapists and other health care professionals about their understanding of self-management and their needs for training about using self-management approaches with PwPMS.

Baseline Assessments.

The questionnaires will measure the impact MS has on functional abilities, including, a range of activities of daily living and quality of life:

1. Modified Fatigue Impact Scale (MFIS)
2. Multiple Sclerosis Impact Scale (MSIS-29)
3. EQ-5D-5L (EuroQol quality of life measure)
4. OX-PAQ (Oxford Participation and Activity Questionnaire)
5. University of Washington self-efficacy scale (UW-SES)
6. Participant Impression of Change (at 3 and 6 months only)

Follow-up. At 3 months post baseline, participants will again complete the above outcome measures, plus the Patients' Global Impression of Change online. Participants will also be telephoned to participate in an interview about their experiences of the intervention.

At 6 months post baseline participants will complete the same questionnaires as previously completed at baseline and 3 months.

Sample size. Twenty-one participants will be recruited to this feasibility study. The sample size is based on the width of a 95% confidence interval for a proportion and allows the proportion of eligible subjects recruited (70%) to be estimated to within +/-20%. The lower 95% confidence interval is 50% which is the minimum acceptable recruitment proportion.

Main analysis. The primary outcome will be based on the feasibility of the study in terms of quantitative measures recruitment, retention and intervention uptake. These proportions will be tabulated with 95% confidence intervals alongside the CONSORT chart which will detail the reasons for exclusion, refusal and dropout. For the clinical secondary outcomes, the data completeness for each measure will be tabulated. The distributions of the outcomes scores will be investigated and appropriate summary measures for the whole group tabulated with 95% confidence intervals at baseline and follow-up time points. An assessment of dropout bias will be made via tabulation of baseline measures for those with complete follow-up data and those who were not followed-up. No formal hypothesis tests will be carried out in the analysis.

Adherence data will be summarised using the following definitions

1. Study adherence: the proportion of participants returning completed outcomes measures
2. Intervention Uptake. Participants will be asked to use the LEAP-MS package during a 3-month period. This is a web-based package and as such participant 'logins' can be monitored. A pre-specified inactivity period of 2 weeks on the website by any one participant will automatically be logged and flagged to the corresponding patients' physiotherapist, who will then contact the participant to offer any further support.

Factors such as disease severity and self-efficacy that may plausibly impact on adherence and retention will be explored with graphical displays.

Progression criteria for a future evaluation will be defined through documentation of adherence and retention as benefits and challenges associated with adherence or lack thereof. We will also assess and record any adverse events that may be reported during participation in the feasibility study and in will consider excessive fatigue or pain that may be related to physical activity.

Qualitative data collection. Interviews with participants and physiotherapists Where consent is provided, interviews will be audio recorded and transcribed verbatim. References to identifiable personal details such as name, address, and date of birth, will be removed from the transcripts.

Observational data Observational data (i.e. proxemic sketches and kinesics data) will be collected on paper Case Report Forms (CRFs) and kept securely in locked files using participant identification (ID) numbers only.

Data from online interaction Data collected from online interaction (emails between patient and physiotherapist, goal setting and activity records) will be also be held on secure Centre for Trials Research (CTR) servers for analysis.

Quality Control and Assurance. The study risk assessment has been used to determine the intensity and focus of central and on-site monitoring activity in the LEAP-MS study. Low monitoring levels will be employed and are fully documented in the Study monitoring plan.

ELIGIBILITY:
Inclusion Criteria:

* People aged 18 and over
* With progressive MS
* Having an Expanded Disability Status Scale (EDSS) score of 6, 6.5, 7, 7.5 or 8.

Exclusion Criteria:

* aged under 18
* an EDSS <6 or >8
* relapsing-remitting or non-progressive MS
* unable to understand written and spoken English
* lacking capacity to consent on their own behalf
* pregnant or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 6 months
  assessed as the percentage of those submitting online permission to contact forms who are eligible and who consent to participation.
  The primary outcome will be based on the feasibility of the study in terms of quantitative measures of recruitment, retention and intervention uptake. These proportions will be tabulated with 95% confidence intervals alongside the CONSORT chart. No formal hypothesis tests will be carried out in the analysis. Intervention uptake data will be summarised based on the proportion of participants engaging with the intervention. Factors such as disease severity (as represented by EDSS scores) and self-efficacy that may plausibly impact on intervention uptake and retention will be explored. Safety data will be collected through self-reporting by the participant on the digital interactive education and activity tool. Acceptability of the intervention to both PwPMS and physiotherapists (usability, content, design, and language) and fidelity will be assessed.
Retention rate | 6 months
  will be measured as the percentage of individuals who complete the 3 and 6 month follow-up assessments
Intervention uptake | 6 months
  will be defined as percentage of intervention sessions completed which may be reflected as number of completed physiotherapy led coaching sessions and number of remote physiotherapist contacts, website log in rates, length of time between each log in episode and duration of logged activity.
Costs associated with intervention delivery | 6 months
  potential therapist travel and contact time will be recorded
Incidence of Treatment-Emergent Adverse Events | 6 months
  will be assessed by an online process of self-reporting by the participant
Acceptability assessment (process evaluation) | 6 months
  will focus on content, design, language and adaptability to personal needs and will be assessed through use of any remote contact facility and semi-structured interviews (either face to face or by telephone) with participants who completed the intervention and physiotherapists who delivered the intervention
Fidelity of intervention delivery | 6 months
  will be assessed through sampled observations of interactive physiotherapy consultations.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Busse, Principal Investigator — Cardiff Unviersity
Locations (1):
- Centre for Trials Research, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Latchem-Hastings J, Randell E, Button K, Jones F, Lowe R, Dawes H, Wood F, Davies F, Poile V, O'Halloran R, Stensland B, Tallantyre E, Playle R, Edwards A, Busse M. Lifestyle, exercise and activity package for people living with progressive multiple sclerosis (LEAP-MS): protocol for a single-arm feasibility study. Pilot Feasibility Stud. 2021 May 22;7(1):111. doi: 10.1186/s40814-021-00852-w. PMID 34022955
- [Derived] Lowe R, Barlow C, Lloyd B, Latchem-Hastings J, Poile V, Scoble C, Dean-Young A, Button K, Playle R, Busse M. Lifestyle, Exercise and Activity Package for People living with Progressive Multiple Sclerosis (LEAP-MS): adaptions during the COVID-19 pandemic and remote delivery for improved efficiency. Trials. 2021 Apr 16;22(1):286. doi: 10.1186/s13063-021-05245-1. PMID 33863342